CLINICAL TRIAL: NCT04846556
Title: Cancer Associated Thrombosis: What is the Proportion of Patients Ineligible to a Study as CARAVAGGIO (a Retrospective Multicenter Study)
Brief Title: Cancer Associated Thrombosis : What is the Proportion of Patients Ineligible to a Study as CARAVAGGIO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN352021/CHUSTE
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Venous Thromboembolism; Cancer
Keywords: Cancer; thrombosis; epidemiology; cancer-associated venous thromboembolism (CAT); venous thromboembolic event
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms; Thrombosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- venous thromboembolic event related to cancer: Patients admitted for a venous thromboembolic event related to their cancer will be included A data collection will be realized. Patients admitted between 2017 and 2019 at Saint-Etienne University Hospital, Louis-Mourier Hospital (AP-HP) and Amiens University Hospital.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection : gender, weight, biological data (platelets, hemoglobin, creatinine, liver function tests), performance status, type of Venous Thromboembolic Event (VTE) and cancer, anticancer and anticoagulant therapy, adverse events (bleeding, recurrence of Venous Thromboembolic Event (VTE), death) up to 6 months after their Venous Thromboembolic Event (VTE).

SUMMARY:
Venous thromboembolism is a common and fatal disease closely related to cancer. The therapeutic challenge is major due to the high risk of recurrent thromboembolism and bleeding in patients with cancer.

Guidelines recommend the use of low molecular-weight heparin for the treatment of Cancer-Associated venous Thromboembolism (CAT) at least for 3 to 6 months of treatment.

However, recent advances through the results of several therapeutic trials such as CARAVAGGIO (NCT03045406) open the door to the use of Direct Oral AntiCoagulants (DOACs) as first-line therapy.

Nevertheless, extrapolation of its results may be limited owing to a large number of inclusion and exclusion criteria, which may have selected a reduced population.

The proportion of patients admitted with acute CAT who may not eligible to a trial as CARAVAGGIO is unknown.

DETAILED DESCRIPTION:
The aim of this study si to assess this proportion in a retrospective multicenter study, of patients admitted for acute Cancer-Associated venous Thromboembolism (CAT).

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients with a newly diagnosed, objectively confirmed:

* symptomatic or unsuspected Deep Vein Thrombosis (DVT) (any location)
* symptomatic or unsuspected Pulmonary Embolism (PE)

Consecutive patients with any type of cancer whose primary brain tumor or known intracerebral metastases and acute leukemia that meets at least one of the following:

* Active cancer defined as diagnosis of cancer within six months or receiving treatment for cancer or any treatment for cancer or recurrent locally advanced or metastatic cancer.
* Cancer diagnosed within 2 years.

Exclusion Criteria:

* pregnant women or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for a venous thromboembolic event related to their cancer will be included between 2017 and 2019 at Saint-Etienne University Hospital, Louis-Mourier Hospital (AP-HP) and Amiens University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of cancer patients with a venous thromboembolic event (VTE) ineligible for CARAVAGGIO study | Up to 6 months after venous thromboembolic event
  Patient having at least one of the following exclusion criteria (from CARAVAGGIO study) :
  * ECOG (Eastern Cooperative Oncology Group ) Performance Status III or IV;
  * life expectancy of less than 6 months;
  * thrombectomy, vena cava filter insertion, or thrombolysis used to manage the index episode;
  * indication for anticoagulant treatment for a disease other than the index VTE episode;
  * thienopyridine therapy (clopidogrel, prasugrel, or ticagrelor) or aspirin over 165 mg daily or dual antiplatelet therapy;
  * recent brain, spinal or ophthalmic surgery
  * hemoglobin level lower than 8 g/dL or platelet count <75x10^9/L or history of heparin induced thrombocytopenia;
  * creatinine clearance < 30 ml /min
  * acute hepatitis, chronic active hepatitis, liver cirrhosis;
  * uncontrolled hypertension;
  * concomitant use of strong inhibitors or inducers of cytochrome;
  * bacterial endocarditis;

SECONDARY OUTCOMES:
Drugs used for their VTE | Up to 6 months after venous thromboembolic event
  Collected in medical history.
Confirmed recurrent Venous Thromboembolic Event (VTE) | Up to 6 months after venous thromboembolic event
  Collected in medical history.
  * Pulmonary embolism
  * deep venous thrombosis
Bleeding event | Up to 6 months after venous thromboembolic event
  Collected in medical history.
Death | Up to 6 months after venous thromboembolic event
  Collected in medical history.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bertoletti, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (3):
- France (3):
  - CHU d'Amiens, Amiens
  - Hôpital Louis Mourier, Colombes
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No